CLINICAL TRIAL: NCT05473845
Title: The Effect of Acupressure and Reiki on Pain and Fatigue Levels in Cancer Patients Receiving Palliative Care
Brief Title: The Effect of Acupressure and Reiki on Pain and Fatigue Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, PhD, MSc, RN, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUTLİ
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Acupressure; Cancer Pain; Fatigue
MeSH Terms: conditions — Cancer Pain; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure (Experimental): Acupressure intervention
  Interventions: Procedure: Acupressure intervention
- Reiki (Experimental): Reiki intervention
  Interventions: Procedure: Reiki intervention
- Control (No Intervention): No intervention.

INTERVENTIONS:
Procedure: Acupressure intervention — Acupressure
  Arms: Acupressure
Procedure: Reiki intervention — Reiki
  Arms: Reiki

SUMMARY:
This research was conducted with the aim of determining the effect of levels of pain and fatigue of acupressure and Reiki application on cancer patients receiving palliative care. The research was a single-blind, repeated measures, randomized controlled study. Research data were collected between February and July 2022. The research sample consisted of acupressure and Reiki application groups and a control group with 52 patients in each group, a total of 156 patients. Data was collected by means of a Patient Description Form, an Analgesic Follow-up Form, the Eastern Cooperative Oncology Group Performance Status Scale, the Numeric Pain Rating Scale, and the Brief Fatigue Inventory.

ELIGIBILITY:
Inclusion Criteria:

1. having a diagnosis of third or fourth-stage cancer,
2. being aged 18 years or older,
3. having had pain for at least one month in connection with cancer treatment or the symptoms of the disease,
4. using NSAII or non-opioid analgesics,
5. having a status of 3 or more on the Numeric Pain Rating Scale (NPRS),
6. having a score of 0-3 on the ECOG-PS scale

Exclusion Criteria:

1. having a diagnosis of first or second-stage cancer,
2. being aged less than 18 years,
3. having bone or brain metastasis,
4. using opioid analgesics,
5. having a status of less than 3 on the NPRS,
6. having a status of between 4 and 5 on the ECOG-PS scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | on the second day of the starting week
  A score of 0 indicates no pain, 1-3 slight pain, 4-6 moderate pain, and 7-10 severe pain .
Brief Fatigue Inventory | on the second day of the starting week
  It is scored between 0 and 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Hediye Utli, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No